CLINICAL TRIAL: NCT01376934
Title: Phase 1 Study of Two Techniques in Hysteroscopy That Compare Carbon Dioxide Versus Saline Solution
Brief Title: Clinical Trial of Hysteroscopy in Postmenopausal Women to Compare Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Departamento de Toco-Ginecologia do CAISM, UNICAMP
Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01/2011/PC
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Postmenopausal Women; Hysteroscopy
Keywords: hysteroscopy; saline solution; carbon dioxide; compare two techniques in office hysteroscopy co2 and saline solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: procedure hysteroscopy — office hysteroscopy with gas or saline solution

SUMMARY:
Nowadays,hysteroscopy is a golden standard procedure to describe the morphology of uterine cavity and investigate of abnormal uterine bleeding . The success of the procedure is based on the distension of the cavity . It can cause pain and discomfort and sometimes the procedure fails. . There are two techniques to make the procedure , one with gas and the other with saline solution. Objective: to compare two techniques concerning pain , procedure duration and image quality

DETAILED DESCRIPTION:
The objective of this study is to compare two techniques in office hysteroscopy.In this clinical trial postmenopausal women will undergo a diagnostic hysteroscopy using carbon dioxide or saline solution to uterine cavity distension.

There will be two groups of 70 women each. The objective is to determine which technique provides better image,time of procedure and less discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Women post-menopausal with abnormal uterine bleeding, ultrasound with thick endometrial distorted

Exclusion Criteria:

* Women with uterine malformations
* Women with mental retardation
* Women underwent pelvic radiotherapy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the comfort in office hysteroscopy | one year
  140 women will undergo office hysteroscopy to evaluate pain, time of the procedure and image quality using two techniques one with gas and the other with saline solution.

CONTACTS AND LOCATIONS:
Overall Officials: Valter Fausto Santos, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Departamento de Tocoginecologia FCM UNICAMP, Campinas, São Paulo, Brazil